CLINICAL TRIAL: NCT06832670
Title: Nursing Strategies to Increase Vaccination Rates in Adolescents: Education, Video Animation and Games
Acronym: Adolescent Vax
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hakan Avan, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: hakanavan-0003
Record Dates: First submitted 2025-02-03; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Health; Vaccination Hesitancy; Adolescent Health
Keywords: Nursing Strategies; Vaccination Rates; Adolescents; Health Education; Video Animation; Health Belief Model; Game-Based Learning
MeSH Terms: conditions — Vaccination Hesitancy; Health Education | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Other: intervention
- control group (Sham Comparator)
  Interventions: Other: active comparator

INTERVENTIONS:
Other: intervention — Participants in the intervention group will receive vaccine education, video animation and game practice.
  Other Names: video animation; game practice; vaccine education; active comparator
  Arms: intervention
Other: active comparator — There will be no intervention in this group. It will continue its active education.
  Arms: control group

SUMMARY:
Purpose: This study aims to evaluate how immunization education, video animation, and game interventions based on the Health Belief Model (HBM) affect the immunization decisions of late adolescents. The findings could contribute to the development of targeted interventions to increase vaccine acceptance among adolescents.

Hypotheses:

Does the educational intervention, video animation, and game application affect adolescents' knowledge of vaccines? Do these interventions influence adolescents' positive attitudes towards vaccines? Will the interventions lead to significant changes in adolescents' health beliefs, especially regarding perceived risks, benefits, and barriers? Do the interventions increase vaccine acceptance and vaccination rates among adolescents? Do the interventions reduce vaccine hesitancy among adolescents? Can the Health Belief Model-based interventions provide an effective communication strategy to increase vaccine acceptance?

Method:

The research will be conducted from March 3 to March 30, 2025. Participants will undergo immunization education, video animation, and game applications. Expert opinions will be consulted for developing educational materials, videos, and games. Institutional approval will be obtained, and an informed consent form will be distributed to participants. Those who volunteer will be assigned numbers, and participants for the intervention and control groups will be selected using simple random sampling.

Interventions:

Educational Material: Aimed at increasing awareness about vaccines, the education focuses on the perceived risks, benefits, and barriers to vaccination.

Video Animation: A video that explains how vaccines work, strengthen the immune system, and address perceived risks and benefits.

Game Application: A simulation game called "infected interaction," where participants learn about the spread of infectious diseases during social interactions.

Inclusion Criteria:

Inclusion: Adolescents aged 18-21, willing to participate, complete research forms, and attend the sessions.

Exclusion: Withdrawal from the study.

Variables:

Independent Variables: Gender, age, income, school, chronic illness, etc. Dependent Variables: Scale scores.

Data Collection Tools:

Adolescent Introductory Questionnaire: A form with 14 questions about demographic information and attitudes toward vaccination.

Vaccine Hesitancy Scale: A 9-item scale measuring vaccine hesitancy. Self-Efficacy Scale: A 23-item scale to assess adolescents' self-efficacy in various contexts.

Statistical Analysis:

Sample size was determined by power analysis: 210 participants (105 intervention, 105 control). Data will be analyzed using IBM SPSS Statistics V 26. Normal distribution will be assessed with the Shapiro-Wilk test, and homogeneity of variance will be tested with Levene's test. Pre- and post-test scores will be compared using repeated measures ANOVA. A p-value of <0.05 will be considered statistically significant.

Expected Outcomes:

Increased Knowledge: It is expected that educational interventions and video animations will improve adolescents' knowledge about vaccines, potentially influencing their attitudes.

Positive Attitude Change: The intervention may lead to more positive attitudes towards vaccination.

Changes in Health Beliefs: The intervention could alter adolescents' perceived risks, benefits, and personal beliefs regarding vaccines.

Increased Vaccine Acceptance: The study may demonstrate that these interventions increase vaccine acceptance and vaccination rates.

Effective Communication Strategies: The study may identify effective communication strategies for increasing vaccine acceptance among adolescents.

Contribution to Public Health: This research could show that interventions targeting adolescents may play a critical role in improving public health by reducing the spread of infectious diseases.

DETAILED DESCRIPTION:
Introduction

The World Health Organization (WHO) defines adolescents as individuals between the ages of 10 and 19, a group that constitutes more than 15% of the global population. Psychosocial maturation during adolescence can be divided into three stages: early adolescence (ages 10-14), middle adolescence (ages 15-17), and late adolescence (ages 18-21).

Although most adolescents are healthy, they account for 6% of the global disease and injury burden. Additionally, risk factors for many adult diseases begin or intensify during adolescence. This highlights the importance of adolescent health as a global priority for individual quality of life, future adult health, and societal well-being. Adolescents are particularly vulnerable to infectious diseases, some of which can be prevented through vaccination.

In both the United States (U.S.) and globally, routine childhood immunizations are among the most effective and cost-efficient public health interventions for preventing infectious diseases and early death. In the U.S., more than 100 million cases of vaccine-preventable diseases, such as measles, mumps, rubella, and pertussis, have been prevented. However, adolescents face increased risks of infectious diseases due to biological, behavioral, and environmental factors, making them an important target group for vaccination programs.

Furthermore, childhood and adolescent vaccinations contribute to reducing many preventable diseases while also providing additional health benefits. For example, the HPV vaccine is responsible for preventing approximately 4.5% (640,000 cases) of new cancer cases worldwide. However, HPV vaccination rates among adolescents remain insufficient compared to other vaccines. Factors such as low parent awareness, concerns about vaccine safety, and fears about vaccination increasing sexual activity are key contributors to this issue. Globally, 13.5 million children miss at least one routine vaccine, leading to approximately 1.5 million deaths from vaccine-preventable diseases. Vaccine hesitancy refers to the delay or refusal of vaccination, despite its availability, which negatively impacts immunization efforts.

Vaccination rates for adolescents, especially for Td, flu, and HPV vaccines, are not at optimal levels. Adolescents are at risk for certain vaccine-preventable diseases due to various age-specific behavioral, environmental, and biological factors. For example, recent outbreaks of invasive meningitis in the U.S. primarily occurred on university campuses, where adolescents and young adults live in close proximity and socialize frequently.

Barriers to immunization include limited time, health systems, competing parental priorities, and vaccine hesitancy. Additionally, communication and educational programs are critical to managing vaccine hesitancy in adolescents. These programs should address not only insufficient vaccination coverage for childhood diseases and waning immunity from early childhood vaccination series but also primary vaccination for diseases that specifically affect adolescents. Successful vaccination strategies for adolescents demonstrate the benefits of vaccination through motivational elements and rewards, using age-appropriate, comprehensive, youth-friendly, and evidence-based information and education.

The Health Belief Model (HBM) is a widely used theory to increase vaccine knowledge and vaccination rates. The HBM consists of components such as perceived susceptibility, perceived severity, perceived benefits, perceived barriers, and self-efficacy. This model provides an important framework for understanding the factors that influence individuals' participation in vaccination programs.

Objective: The purpose of this study is to assess how vaccination education, video animation, and game applications, based on the components of the Health Belief Model, affect late adolescents' vaccination decisions. The findings can contribute to the development of targeted interventions to increase vaccine acceptance among adolescents. The importance of vaccination and effective communication strategies play a critical role in achieving adolescent and public health goals.

Research Hypotheses:

1. Hypothesis 1: Does the education intervention, video animation, and game application have an impact on adolescents' knowledge level about vaccines?
2. Hypothesis 2: Does the education intervention, video animation, and game application influence adolescents' positive attitudes toward vaccines?
3. Hypothesis 3: Does the education intervention, video animation, and game application lead to significant changes in adolescents' health beliefs, particularly perceived risks, benefits, and barriers?
4. Hypothesis 4: Does the education intervention, video animation, and game application increase adolescents' vaccination decisions and vaccination rates?
5. Hypothesis 5: Does the education intervention, video animation, and game application reduce vaccine hesitancy among adolescents?
6. Hypothesis 6: Based on the Health Belief Model, does the education intervention, video animation, and game application provide an effective communication strategy for adolescents and increase vaccine acceptance? Method Research Model: The research will be conducted between March 3-30, 2025. Participants will undergo vaccination education, video animation, and game application. Expert opinions will be sought for the development of educational materials, video animation, and game applications. Institutional permission will be obtained, and informed consent forms will be distributed to the participants. Volunteers will be assigned a number, and participants for the intervention and control groups will be selected through simple random sampling. The research will be conducted in three sessions. In the first session, a pre-test will be administered to the group participating in the study ("Adolescent Introduction Questionnaire," "Vaccine Hesitancy Scale (VHS)," and "Self-Efficacy Scale (SES)"). Following this, the researcher will provide education on vaccines. This session will take approximately 30-35 minutes, including the administration of the questionnaires. One week after the first session, the second session will be scheduled. In the second session, a video animation will be presented, lasting about 4-6 minutes. After a 15-minute break, the third session will be held, during which the "infected interaction" game will be played, followed by post-test questionnaires.

The control group will also complete the pre-test on the same day but in a different environment from the intervention group. The control group will continue with their routine training, and on the day the intervention group's post-test is administered, the same questionnaires will be applied to the control group. The data collection process will take about 10-15 minutes. After the research is completed, the control group participants will receive the same vaccination education, video animation, and game application.

Education Material Application: In this research, participants are provided with educational material based on the components of the Health Belief Model (HBM). The material is designed to increase vaccination rates and raise awareness among participants about vaccines. The content is structured around key HBM components, such as perceived susceptibility, perceived severity, perceived benefits, perceived barriers, and self-efficacy.

The educational material aims to inform participants about the risks, benefits, and potential barriers related to vaccination, helping them become more informed about the factors influencing their vaccination decisions. This education is designed to positively influence participants' vaccine acceptance and general attitudes toward vaccines.

Video Animation Application: Participants in this study will be shown a video animation aimed at increasing knowledge and awareness about vaccines. The animation's goal is to explain how vaccines work, how they strengthen the immune system, and to provide information on perceived risks, benefits, and barriers related to vaccination.

The animation will cover topics such as how vaccines affect the body, contribute to the immune system, and influence vaccination decisions. The animation will be about 4 minutes long and will help participants increase their knowledge of vaccines and develop more informed attitudes toward vaccination.

Game Application: Participants will play an "infected interaction" game designed to simulate social interactions and the spread of infectious diseases. The goal of the game is for participants to observe how infected individuals make contact with others and the impact of these interactions on disease transmission.

During the game, two participants will secretly be marked as "infected." These infected individuals will be indicated with a symbol or sign known only to them. The participants will then be asked to socialize freely with others in the group for two minutes. During this interaction, the infected participants will secretly pass on the infection signal to other participants they come into contact with. After the 2-minute interaction, researchers will calculate which participants were infected and whether the infection was passed on to others.

Variables: Independent Variables: Gender, Age, Income Level, School, Presence of Chronic Diseases, etc. Dependent Variables: Scale scores

Data Sources: The following tools will be used to collect data:

* "Adolescent Introduction Questionnaire" containing 14 questions on socio-demographic characteristics and vaccine-related topics
* "Vaccine Hesitancy Scale (VHS)" developed by the SAGE working group and validated by Shapiro et al. (2018) to measure hesitancy toward childhood vaccines
* "Self-Efficacy Scale (SES)" developed by Sherer and Maddux (1982) and adapted into Turkish by Gözüm and Aksayan (1999) to measure general self-efficacy perceptions Statistical Analysis of the Study: Sample Size Calculation Method: Based on Power Analysis (two-tailed hypothesis, 5% significance level, 95% power, 0.5 medium effect size), the sample size will be 210 participants (105 in the control group and 105 in the intervention group).

Comparison Groups and Analytical Methods: Data will be analyzed using IBM SPSS Statistics Standard Concurrent User V 26. The normality of numerical variables will be tested using the Shapiro-Wilk test, and homogeneity of variances will be tested using the Levene test. Independent samples t-tests will be used to compare BMI values between groups. Fisher's exact test will be used to compare categorical variables. Paired sample t-tests will be applied to compare pre- and post-test scale scores, and Bonferroni correction will be applied in the analysis of main effects. p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-21
* Willing to participate in the research
* Completes all research forms
* Fully participates in the training sessions

Exclusion Criteria:

* Desire to withdraw from the research

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
1. Increase in Vaccine Knowledge and Positive Attitude Change Toward Vaccines | 3 weeks
  The video animation, game application and educational program are expected to increase adolescents' knowledge about vaccines. This increased knowledge may lead to changes in attitudes towards vaccines and general health beliefs.
  The "Vaccine Hesitancy Scale" will be used for evaluation. The score obtained from the scale and its subdimensions is calculated by summing the points from the relevant items, and an increase in the score indicates a decrease in vaccine hesitancy. Although there is no specific cutoff point for the scale, the total score can range from 9 to 45 points.
2. Increase in Vaccination Acceptance Rates and Contribution to Public Health | 3 weeks
  This study may show that video animation, game implementation and educational interventions increase adolescents' vaccine acceptance, which may be valuable for the development of future public health strategies. The "Self-Afficacy-Efficacy Scale" will be used for the assessment. A score between 23 and 115 can be obtained from the scale. A higher score indicates a higher perception of Self-Efficacy-Competence regarding vaccines. The scale consists of four sub-dimensions.

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected, all IPD underlying the results in a publication
Supporting Information: Study Protocol